CLINICAL TRIAL: NCT04528433
Title: A Randomized Controlled Study of Medical-education-community Collaborated Intervention in Children With Attention Deficit Hyperactivity Disorder
Brief Title: A Randomized Controlled Study of Medical-education-community Collaborated Intervention in Children With ADHD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xlklmy01
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The present study will be carried out using a parallel randomized study design. Each participant will be randomly assigned either to the collaborated intervention or to the routine clinical care control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The medical treatment of participants will be given by a doctor who does not know the study group of the patient. The investigator of the primary outcome and secondary outcome will also be unaware of the grouping of the patient. One psychiatrist blind of grouping will ask parents about the ADHD symptom of their children and rate it with SNAP-IV score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical-education-community Collaborated Intervention (Experimental)
  Interventions: Behavioral: Medical-education-community Collaborated Intervention
- routine clinical care (Active Comparator)
  Interventions: Behavioral: routine clinical care

INTERVENTIONS:
Behavioral: Medical-education-community Collaborated Intervention — The Medical-education-community Collaborated Intervention adds an additional part in comparison with the control group of classroom management guidance for teachers, review and practice organizational skills based on school daily activities in the school, teacher rewards and encouragement of students.
  Arms: Medical-education-community Collaborated Intervention
Behavioral: routine clinical care — Routine clinical care includes a structured family behavioral intervention for ADHD symptom management and organizational skill training, the medication will be used if necessary.
  Arms: routine clinical care

SUMMARY:
This study is designed to test if the medical-education-community collaborated intervention can reduce the symptoms of children with Attention deficit hyperactivity disorder (ADHD) compared to routine clinical care. Investigators will also evaluate if the intervention will positively affect organizational skills and academic achievement compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ADHD
* Doctor rated SNAP-IV Inattention of Hyperactivity/Impulsivity score>12
* Full-Scale Intelligence Quotient>=80 (Wechsler intelligence scale for children-IV)

Exclusion Criteria:

* Accepting any type of psychological treatment during the intervention
* Comorbid with epileptic disorder or other existing physical disorder, Tourette syndrome, Autism Spectrum Disorder, learning disorder, mood disorder, psychiatric disorder, or under suicidal risk
* Attending any other clinical research at the same time

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
total score change in SNAP-IV scale | Baseline, 3 months after enrollment
  It is a repeated measurement. The Swanson, Nolan, and Pelham Questionnaire (SNAP-IV) Rating Scale is a revised version of the Swanson, Nolan and Pelham (SNAP) Questionnaire that utilizes the DSM-IV criteria for ADHD and oppositional defiant disorder, rated by caregiver or professionals. It comprises three subscales: Inattention, Hyperactivity/Impulsivity, and Oppositional Defiant Disorder. The score of each item is rated with a 4-point Likert scale (0 = not at all, 3 = very much). We choose the total score ofInattention and Hyperactivity/Impulsivityfor the evaluation of change in ADHD symptom in children. The score is calculated by adding all the items inthe two subscales. The change of score is calculated by score at 3 months enrollment minus score at baseline (enrollment).

SECONDARY OUTCOMES:
total score change in Behavior Rating Inventory of Executive Function scale | Baseline, 3 months after enrollment
  It is a repeated measurement. The Behavior Rating Inventory of Executive Function(BRIEF) Scale reflects the performance of children's deficits in executive function in daily life, which covers a number of organizational skills involved in organizational skills training. We choose the total score ofBRIEF for the evaluation of change in organizational skills in children. The score is calculated by the published recording chart. The change of score is calculated by score at 3 months enrollment minus score at baseline (enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Mengyao Li, PhD, Study Chair — Department of Psychological Medicine, Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: Undecided